CLINICAL TRIAL: NCT03276299
Title: Learning and Encouragement Effect on 6 Minute Walking Test in Children Between 6 and 12 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Child6MWT
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Healthy Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- test 1 (Active Comparator): six minute walking test
  Interventions: Other: six minute walking test
- test 2 (Experimental): six minute walking test
  Interventions: Other: six minute walking test
- test with encouragement (Experimental): six minute walking test
  Interventions: Other: six minute walking test
- test without encouragement (Active Comparator): six minute walking test
  Interventions: Other: six minute walking test

INTERVENTIONS:
Other: six minute walking test — six minute walking test
  Arms: test 1; test 2; test without encouragement
Other: six minute walking test — six minute walking test with encouragement
  Arms: test with encouragement

SUMMARY:
Evaluation of the learning and encouragement effect on six minutes walking test in children under 12 years

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* acute or chronic lung, cardiac or neuromuscular disease
* at risk of- or overweight (BMI higher than 85th percentile for children of the same age and sex)
* a motor disability

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
distance | six minutes
  walked distance

SECONDARY OUTCOMES:
heart rate | six minutes
  heart rate
pulsed oxygen saturation | six minutes
  pulsed oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique universitaire Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morales Mestre N, Audag N, Caty G, Reychler G. Learning and Encouragement Effects on Six-Minute Walking Test in Children. J Pediatr. 2018 Jul;198:98-103. doi: 10.1016/j.jpeds.2018.02.073. Epub 2018 Apr 24. PMID 29703575